CLINICAL TRIAL: NCT06740539
Title: Atrial Fibrillation with Heart Failure with Preserved Ejection Fraction: Treatment Strategies-Catheter Ablation Vs. Anti-Atrial Arrhythmia Drugs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: The Third Affiliated Hospital of Anhui Medical University (Unknown); Hefei Second People's Hospital (Unknown); The Second People's Hospital of Anhui Province (Other); Hefei Binhu Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, Professor, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPHF-AF
Record Dates: First submitted 2024-12-15; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: HFpEF - Heart Failure with Preserved Ejection Fraction; Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ablation Group (Experimental): Ablation Group: Received heart failure treatment combined with ablation
  Interventions: Procedure: Catheter ablation of atrial fibrillation
- Drug Control Group (No Intervention): Received heart failure treatment combined with heart rate control.

INTERVENTIONS:
Procedure: Catheter ablation of atrial fibrillation — Catheter ablation of atrial fibrillation
  Arms: Ablation Group

SUMMARY:
A comparison of whether catheter ablation improves the prognosis (all-cause mortality and/or the composite endpoint of MACE) and reduces the recurrence rate of atrial fibrillation (AF) in patients with AF and heart failure with preserved ejection fraction (HFpEF), compared to anti-atrial arrhythmia drugs (AAD). This trial was randomly divided into two groups: the anti-AAD drug group and the catheter ablation group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* The patient is willing and able to comply with the protocol and has provided written informed consent.
* Paroxysmal or persistent atrial fibrillation (AF).（Persistent AF was defined as AF which is sustained beyond 7 days, or lasting less than seven days but necessitating pharmacologic or electric cardioversion. Included within the category of persistent AF is 'long-standing persistent AF', defined as continuous AF of >1-year duration. AF episodes had to be documented in the last 3 months prior to enrollment by ECG, Holter ECG, Loop Recorder, memory of the implanted device (ICD/CRT-D), or any other suitable device.）
* Failure or intolerance of antiarrhythmic drug therapy or unwillingness to take antiarrhythmic drugs.
* Diagnosed with Heart Failure with Preserved Ejection Fraction (HFpEF).（(1) a history of hospitalization for HF with symptoms classified as New York Heart Association (NYHA) class II, III, or IV; (2) LVEF ≥ 50%; (3) at least one of the following cardiac structural abnormalities identified by echocardiography: left ventricular hypertrophy, left atrial enlargement, or diastolic dysfunction; and (4) elevated levels of N-terminal pro-brain natriuretic peptide (NT-proBNP), with a threshold of ≥400 pg/mL for pa-tients with SR at admission and ≥600 pg/mL for patients with AF at admis-sion.)
* New York Heart Association class II, III, or IV.

Exclusion Criteria:

* Previous left heart ablation procedure for AF.
* Contraindication to chronic anticoagulation therapy or heparin.
* Documented left atrial diameter >6 cm, optimally from the parasternal long-axis view.
* Acute coronary syndrome, cardiac surgery, angioplasty, or cerebrovascular accident within 2 months prior to enrollment.
* Planned cardiovascular intervention.
* Listed for heart transplant.
* Cardiac assist device implanted.
* Life expectancy ≤ 12 months.
* Mental or physical inability to participate in the study.
* Requirement for dialysis due to terminal renal failure.
* Woman currently pregnant or breastfeeding or not using reliable contraceptive measures during fertility age.
* Enrollment in another investigational drug or device study, or participation in another telemonitoring concept.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2024-12-16 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint was a composite of all-cause death or rehospitalization for worsening HF. | During regular follow-up visits at 3, 6, 12, 24months.
  The primary endpoint was a composite of all-cause death or rehospitalization for worsening HF.

SECONDARY OUTCOMES:
All-Cause Mortality | During regular follow-up visits at 3, 6, 12, 24months.
  All deaths and all heart transplants because of terminal heart failure (HF) will be included.
Worsening of Heart Failure Requiring Unplanned Hospitalization | During regular follow-up visits at 3, 6, 12, 24months.
  Patients requiring intravenous medication for HF (including diuretics, vasodilators or inotropic agents) or a substantial increase in oral diuretic therapy for HF (i.e., an increase of furosemide ≥40 mg or equivalent, or the addition of a thiazide to a loop diuretic) will be deemed to have worsening of HF. Further, rales and/or S3 sound, chest x-ray, worsening of dyspnea, worsening of peripheral edema and increase of New York Heart Association class will be assessed for determination of worsening of HF.Unplanned hospitalization is defined as any in-hospital stay over one date change, and not planned by the Investigator.
Cardiovascular Mortality | During regular follow-up visits at 3, 6, 12, 24months.
  All deaths due to cardiovascular reasons and all heart transplants because of terminal HF. Deaths due to worsening of HF, acute coronary syndrome, cerebrovascular accidents, or other cardiovascular events will qualify for this secondary end point.
Unplanned Hospitalization due to Cardiovascular Reason | During regular follow-up visits at 3, 6, 12, 24months.
  Any in-hospital stay over one date change due to cardiovascular reason, which includes worsening of HF, acute coronary syndrome, cerebrovascular accidents, or other cardiovascular events, and not planned by the Investigator. In case the hospitalization is classified as planned by the Investigator, and the time interval between the decision to hospitalize and the hospitalization is less than 24 hours, the End Point and Adverse Event Committee will give final classification concerning planned or unplanned.
All-Cause Hospitalization | During regular follow-up visits at 3, 6, 12, 24months.
  Any in-hospital stay over one date change.
Cerebrovascular Accident | During regular follow-up visits at 3, 6, 12, 24months.
  Cerebrovascular accident, ischemic or hemorrhagic, describes a clinical and neurological syndrome, based on an acute damage of the brain. The common denominator is the sudden onset of a neurological deficit.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No